CLINICAL TRIAL: NCT00250302
Title: Autologous Implantation of Mesenchymal Stem Cells for the Treatment of Distal Tibial Fractures
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMSC-01-HMO-CTIL
Record Dates: First submitted 2005-11-06; First posted 2005-11-08 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2010-10

CONDITIONS: Tibial Fracture
MeSH Terms: conditions — Tibial Fractures

INTERVENTIONS:
Procedure: autologous mesenchymal stem cells implantation

SUMMARY:
Mesenchymal stem cells are found in bone marrow, and have the ability to differentiate into different tissue types. The primary objective of the study is to examine the safety of using such cells to treat patients suffering from distal tibial shaft fractures. The cells will be isolated from the patient's bone marrow, loaded onto a carrier and implanted locally at the fracture site.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and 65. males not involved in active military duty. females- non child bearing potential. distal tibia third fracture without joint involvement. fracture treated by IM nail, percutaneous plating or external fixation.

Exclusion Criteria:

* active systemic or local infection. history of malignancy radiotherapy or chemotherapy. active autoimmune disease. any past or present immunosuppressive treatment. fracture treated by open reduction. fracture grade gustillo grade IIIB, IIC. use of steroids in past 6 months. chronic renal insufficiency. administration of marrow suppressive drugs. history of metabolic bone disease. administration of drugs that may interfere with bone metabolism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety
Number of patients reaching clinical union of fracture

CONTACTS AND LOCATIONS:
Overall Officials: Meir Liebergall, Prof., Principal Investigator — Hadassah Medical Organization; Rami Mosheiff, Prof., Study Director — Hadassah Medical Organization; Dan Gazit, Prof., Study Chair — Hebrew University
Locations (1):
- Hadassah Medical Organizaton, Jerusalem, Israel